CLINICAL TRIAL: NCT02448602
Title: Scheme Optimization of Acupoints Compatibility and Influence Factors of the Effect
Brief Title: Different Acupoints Compatibility Difference of the Effect of Treatment of the Primary Insomnia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun University of Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); Hengyang Traditional Chinese Medicine Hospital (Other); Second People's Hospital of Hunan (Other); Jilin University (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Tie Li, 973 project management deputy director of the office, Changchun University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChangchunUCM
Record Dates: First submitted 2015-04-14; First posted 2015-05-19 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Primary Insomnia
Keywords: Different acupoints compatibility
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single point group (Shenmen) (Other): Patients will be acupuncture with Shenmen(HT7).
  Interventions: Other: acupuncture
- Sancai coordinated points group (Other): Patients in Sancai coordinated points group, will be acupuncture with Baihui(DU20), Shenmen(HT7), Sanyinjiao(SP6).
  Interventions: Other: acupuncture
- Control group (Other): Patients in Control group, will be acupuncture with at the junction of deltoid and biceps.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Patients will be treated with Shenmen(HT7), needle 1 times a day, 30 min/time, 5 days for a period of treatment, the treatment interval for two days, five intervention treatment, follow-up after 4 weeks.
  Arms: Single point group (Shenmen)
Other: acupuncture — Patients in Sancai coordinated points group, will be treated with Baihui(DU20), Shenmen(HT7), Sanyinjiao(SP6), needle 1 times a day, 30 min/time, 5 days for a period of treatment, the treatment interval for two days, five intervention treatment, follow-up after 4 weeks.
  Arms: Sancai coordinated points group
Other: acupuncture — Patients in Control group, will be treated with at the junction of deltoid and biceps, needle 1 times a day, 30 min/time, 5 days for a period of treatment, the treatment interval for two days, five intervention treatment, follow-up after 4 weeks.
  Arms: Control group

SUMMARY:
With primary insomnia as the research object, by the method of multi-center RCT and needle single cavity and different acupoints compatibility treatment for primary insomnia, to Pittsburgh sleep quality index(PSQI) and evaluation, sleep log evaluation and Polysomnogram(PSG) as the means, such as the single cavity with different acupoints compatibility evaluate clinical curative effect of treating primary insomnia.

DETAILED DESCRIPTION:
In order to establish a spectrum of acupoints compatibility of the law, is clear about the factors affecting the compatibility effect of acupoints, the formation of strong operability of acupoints compatibility optimization evaluation method, the project choice of the clinical acupuncture and moxibustion have curative effect of primary insomnia as the breakthrough point of the study, carried out clinical multi-center RCT research, through objective and scientific evaluation method, comparing the effect of different acupoints compatibility.

Primary insomnia in clinical common disease, frequently-occurring disease, acupuncture curative effect is distinct, disease diagnosis, curative effect evaluation standard. Previous clinical data also show that the primary insomnia is acupuncture clinical diseases. This project by primary insomnia as the research object, research to better guide clinical practice, improve the clinical curative effect, promote acupuncture of the inheritance and innovation, promote scientification of acupuncture and moxibustion, modernization and internationalization, and will have broad prospect of application and significant scientific research value.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Insomnia 's Disease;
* Aged 18-60 (including 18 and 60);
* Does not attend other clinical researchers;
* Participation in the researchers signed informed consent and voluntary;
* Pittsburgh sleep index (PSQI) index > 7 points;
* Athens scale or 6 points;
* Depression scale and anxiety scale 50 points or less.

Exclusion Criteria:

* Breathing-Related Sleep disorder;
* Circadian rhythm disorders;
* Sleep disorders;
* Drug-induced insomnia (such as drug abuse, drug treatment);
* Sleep disorders caused by poor diet, lifestyle factors(Long-term excessive drinking, coffee, tea, etc.);
* All systemic diseases (such as pain, fever, cough, surgery, etc.) and the external environment disturbance factors;
* With cardiovascular, lung, liver, kidney and hematopoietic system such as serious primary diseases;
* Patients with mental illness;
* Pregnancy or breast-feeding women;
* Acupoints with severe skin infections;
* Patients who are afraid of acupuncture;
* Advanced malignant tumor or other serious wasting disease, infection and bleeding;
* Who do not meet the inclusion criteria, poor compliance, treatment, not according to stipulations can not judge the curative effect or data not congruent affect curative effect and safety of judgment;
* Caused by excessive anxiety and depression of patients with insomnia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 333 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index(PSQI) | 9 weeks

SECONDARY OUTCOMES:
Test GABA,Glu,5-HT,Ach,NE,DA in the human brain to reflect the state of brain function by the Encephalofluctuograph(ET) | 5 weeks
Change in Total Sleep Time Measured by PSG | 5 weeks
  Measuring indexes including total record time(TRT), sleep time(SPT), total sleep time(TST, sleep efficiency, sleep latency(SL), sleep cycle changes, awakening times, fall asleep after waking hours, REM times incubation period, incubation period of REM, REM (except the awakening times).
Sleep diary | 5 weeks
Athens insomnia scale | 9 weeks
Self-rating anxiety scale(SAS) | 1 week
Self-Rating Depression Scale(SDS) | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Fuchun Wang, master, Study Chair — Dean
Locations (1):
- The Affiliated Hospital To Changchun University of Chinese Medicine, Changchun, Jilin, China

REFERENCES:
- [Derived] Ha L, Liu X, Liu Y, Zhi M, Jiang H, Zhao J, Wang Y, Xu X, Guo L, Cao J, Chen L, Yuan Y, Li T, Wang F. Scheme optimization of acupoints compatibility and influence factors of the effect. Medicine (Baltimore). 2021 Dec 17;100(50):e27883. doi: 10.1097/MD.0000000000027883. PMID 34918637
- [Derived] Shi XH, Wang YK, Li T, Liu HY, Wang XT, Wang ZH, Mang J, Xu ZX. Gender-related difference in altered fractional amplitude of low-frequency fluctuations after electroacupuncture on primary insomnia patients: A resting-state fMRI study. Brain Behav. 2021 Jan;11(1):e01927. doi: 10.1002/brb3.1927. Epub 2020 Nov 4. PMID 33146953
- [Derived] Wang YK, Li T, Ha LJ, Lv ZW, Wang FC, Wang ZH, Mang J, Xu ZX. Effectiveness and cerebral responses of multi-points acupuncture for primary insomnia: a preliminary randomized clinical trial and fMRI study. BMC Complement Med Ther. 2020 Aug 17;20(1):254. doi: 10.1186/s12906-020-02969-6. PMID 32807158